CLINICAL TRIAL: NCT00849641
Title: Muscle Tissue Oxygenation in Patients With Decompensated Liver Cirrhosis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Regensburg (Other)
Responsible Party: Dr. Sylvia Siebig, MD, University of Regensburg, Germany
Other Study IDs: UR-ST9201/09
Record Dates: First submitted 2009-02-20; First posted 2009-02-24 (Estimated); Last update posted 2009-02-24 (Estimated); Status verified 2009-02

CONDITIONS: Liver Cirrhosis
Keywords: decompensation; septic shock; tissue oxygenation; near infrared spectroscopy
MeSH Terms: conditions — Liver Cirrhosis; Shock, Septic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- 1: patients with decompensated liver cirrhosis admitted to the medical ICU
- 2: critically ill patients without liver cirrhosis, matched to group 1
- 3: healthy control group

SUMMARY:
Patients with decompensated liver cirrhosis exhibit numerous hemodynamic and microvascular changes, i.e., low systemic blood pressure and peripheral vasodilatation. In addition, alterations of tissue oxygenation are described in these patients.

Near-infrared spectroscopy (NIRS) has been proposed as a tool to quantify microvascular dysfunction, for example in patients with sepsis (1) or after trauma (2). NIRS is a non-invasive technique that uses the differential absorption properties of oxygenated and desoxygenated hemoglobin to evaluate skeletal muscle oxygenation (3).

Up to the investigators' knowledge no data exist on NIRS measurements in patients with decompensated liver cirrhosis.

Aims of this study are to evaluate:

* Are there any changes in NIRS parameters in patients with decompensated liver cirrhosis in comparison to other critically ill patients (matched to SAPS II Score) or healthy individuals?
* Is there a correlation with common accepted prognostic scores (MELD Score or indocyanin green clearance) in decompensated liver cirrhosis patients and initial NIRS parameters?
* Does the NIRS trend within the first three days of ICU care in decompensated liver cirrhosis patients receiving fluid replacement therapy correlate with the course of disease?

  1. De Backer D, Creteur J, Preiser JC, Dubois MJ, Vincent JL. Microvascular blood flow is altered in patients with sepsis. Am J Respir Crit Care Med. 2002 Jul 1;166(1):98-104.
  2. Creteur J. Muscle StO2 in critically ill patients. Curr Opin Crit Care. 2008 Jun;14(3):361-6.
  3. Creteur J, Carollo T, Soldati G, Buchele G, De Backer D, Vincent JL. The prognostic value of muscle StO2 in septic patients. Intensive Care Med. 2007 Sep;33(9):1549-56.

DETAILED DESCRIPTION:
Patients fulfilling inclusion criteria and without exclusion criteria will be monitored by NIRS using InSpectra™ technology (Hutchinson, USA) for the first three days of their ICU hospitalization. Besides registration of the NIRS parameters (tissue hemoglobin saturation (StO2), total tissue hemoglobin (THI), dynamic test values by using occlusion testing) baseline characteristics (age, sex, SAPS II Score et.), disease relevant information (etiology of liver cirrhosis, cause of ICU hospitalization) and ICU data (catecholamine therapy, mechanical ventilation, hemodynamic monitoring, fluid therapy) will be recorded. Within the observation time, an indocyanin green-clearance measurement and further laboratory testing will be performed on a daily basis. Data will be pseudonymized and kept confidential according to the guidelines of the local ethics committee.

ELIGIBILITY:
Inclusion Criteria:

* patients with decompensated liver cirrhosis admitted to the medical ICU
* written informed consent signed by the patients or his/her closest family member
* age ≥ 18year

Exclusion Criteria:

* no written informed consent signed by the patients or his/her closest family member

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with decompensated liver cirrhosis
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2009-03; Primary Completion 2010-10 (Estimated); Study Completion 2011-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Sylvia Siebig, MD, Principal Investigator — University of Regensburg
Locations (1):
- University Hospital of Regensburg, Regensburg, Germany